CLINICAL TRIAL: NCT01410708
Title: A Pre-Surgical Study to Evaluate Molecular Changes That Occur in Human Breast Cancer Tissue After Short Term Exposure to Dasatinib and To Correlate These Alterations With Pharmacokinetics Parameters
Brief Title: TORI 104 Pre-Surgical Dasatinib
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-1-0103; TORI 104
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Human Breast Cancer Tissue; Dasatinin
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dasatinib

SUMMARY:
This study will examine the anti-tumor activity, safety and tolerability of dasatinib in adjuvant breast cancer patients in a pre-surgical setting.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the molecular changes which occur in human breast cancer tissue after short-term exposure to dasatinib.

Secondary Objectives:

" To evaluate the molecular effects of short term dasatinib exposure in peripheral blood and on SRC (an oncogene) and EPHA2 signaling pathways in non-tumor cells (peripheral blood).

" To correlate the pharmacokinetic parameters with molecular changes detected in breast cancer tissues and peripheral blood " To evaluate the tolerability and safety of short-term exposure to daily dose of 100 mg twice daily of dasatinib administration

Study Design:

Eligible patients will be registered to receive dasatinib 100 mg orally twice daily starting within 8 days from the time of registration and continuing to the time of the definitive surgery.

Duration of Treatment " No more than 8 days should elapse from the time of registration to the time of the first dose of dasatinib " No more than 28 days should elapse from the time of the initial diagnosis to the time of the first dose of dasatinib " Minimum duration of treatment with dasatinib is 14 days with a minimum of 10 consecutive days of treatment immediately prior to the definitive surgery " Dasatinib shall be administered until the day prior to the definitive surgery " No more than 45 days should elapse from the time of the initial diagnosis to the time of the definitive surgery i.e. maximum duration of treatment with dasatinib is 45 days.

Core Biopsies: Tumor sample must be collected at the time of the initial diagnosis (or in a subsequent procedure) either by core needle or incisional biopsy. Excisional biopsy will not be allowed. A minimum of 4 core biopsies (or the equivalent with an incisional biopsy) is required to perform the molecular analyses. Once the core biopsies have been removed, the samples must be immediately snap-frozen, then stored in liquid nitrogen or at -70 to -80 C at the site. Samples will be shipped to the UCLA laboratory within 30 days of collection.

Tumor Tissue at the time of Definitive Surgery: A second tumor sample (post-dasatinib) must be collected at the time of the patient's surgery in the same manner as above.

Unstained paraffin slides: While most analyses will be performed on the frozen tissue, some molecular testing may require paraffin embedded tissue. The pathology department will be asked to send 4, 5 micron thick, unstained paraffin slides of each the pretreatment (diagnosis biopsy) and from the definitive surgery (8 slides in total) Definitive Surgery: The type of definitive surgery performed will be according to the institution's guidelines. In the event that a sentinel node biopsy procedure is performed, the dye can be injected into the tumor bed after tumor removal. The dye should not be injected into the tumor itself as this may alter the tissue and affect the molecular analyses.

Pharmacokinetic plasma samples and peripheral blood mononuclear cells samples will be collected at the following time points (5 samples each):

1. Baseline, prior to the first dose of dasatinib. Timing of collection: anytime between registration and the first dose of dasatinib.
2. Last day of dasatinib (= on the day prior to surgery) Timing of Collection: patient should be asked to come into the clinic before taking her last morning dose of dasatinib. Blood can be drawn immediately prior to her taking the tablet in the clinic.
3. Last day of dasatinib (= on the day prior to surgery) Timing of Collection: 2-3 hours after the last morning dose
4. Last day of dasatinib (= on the day prior to surgery) Timing of Collection: 6-8m hours after the last morning dose
5. On the day of surgery Timing of Collection: as close as possible to the surgery (+/- 1 hour) Patients will be requested to document the date and time of each dose consumed as well as any details concerning a drug holiday in the patient diary.

Samples from all patients are required to all for the relatively large variability in dasatinib pharmacokinetics (interpatient coefficient of variation is approximately 65 %) The samples will be centrifuged, processed, and shipped. Results from the pharmacokinetics analysis will be correlated with the molecular data.

Number of Patients: 60 evaluable patients

Statistical Analysis:

The primary objective of this trial is to evaluate molecular changes occurring in breast cancer tissue following short-term dasatinib administration. Based on pre-clinical data supporting the role of Src in "triple-negative" breast cancer, the study will aim for 50% of evaluable patients be of this subtype defined as being negative for ER, PR, and HER2 amplification. In cases where HER2 amplification is not determined by FISH at diagnosis, HER2 staining by IHC of 0 or 1+ will be considered negative for enrolment purposes. After 30, 40, and 50 evaluable patients have been accrued, enrolment may be adjusted to reach the goal of 30 triple-negative patients.

Descriptive statistics will be used to compare the pre- and post-treatment molecular findings. A statistical Analysis Plan (SAO) will be finalized at the latest prior to database lock and the analysis details will be provided in the SAP. Descriptive statistics will be used to describe the incidence of adverse events and toxicity, as well as the number of patients in who the study medication was permanently stopped.

Stopping Rules:

Enrolment is completed according to protocol planned sample size, and assessments and requirements are completed as per protocol, the stated objectives of the trial are achieved, recommendation by DMC. Patients may withdraw from the trial at any time at their own request, or they may be withdrawn at any time at the discretion of the investigator or sponsor if continuation of the study would be detrimental to the patient's well being, such as objective disease progression, unacceptable toxicity, noncompliance, second primary malignancy, or logistical considerations

ELIGIBILITY:
Inclusion Criteria:

* Informed signed consent, female, over 18 years of age nad Karnofsky performance status index greater than 80%.
* Histologically proven invasive breast cancer through either core needle biopsy or an incisional biopsy. Excisional biopsy not allowed.
* Tumor must be confined to either the breast or to the breast and ipsilateral axilla. Tumor size of greater than 2cm (T1 with T=2m, T2-T3. Patient can have clinically positive (N1) or clinically negative)
* Neutrophils greater than 1.5 x 109/L, Platelets greater tahn 100 x 109/L, Hemoglobin greater than 10g/dL.
* Total bilirubin less than 1 UNL, AST and ALT less than 2.5 UNL, Alk phos less than 5 UNL, creatinine less than 175umol/L (2mg/dL)
* not more than 28 days from the time of the initial diagnosis and 8 days from registration to the first dose of dasatinib shall elapse.
* Patients must be accessible for treatment and the 30-day follow-up and compliant with study procedures.
* Negative pregnancy test within 7 days prior to registration for women of childbearing potential.

Exclusion Criteria:

* Prior or concurrent systemic anticancer therapy
* Prior or concurrent ipsilateral radiation therapy for invasive or noninvasive breast cancer.
* Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment.
* Any T1 (with exception of T1 with T=2cm) or T4 or N2 or known N3 or M1 breast cancer.
* Concurrent or congestive heart failure, unstable angina pectoris or MI in past 6 months; uncontrolled hypertension or high risk uncontrolled arrhythmias; any history of significant ventricular arrhythmia.
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding of informed consent; active uncontrolled infection.
* Past or prior history of neoplasm other than breast carcinoma, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated.
* Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment should be stopped at least 2 weeks prior to registration.
* Concurrent treatment with other experimental drugs or treatment wih investigational drugs with 30 days of registration.
* Prior hormonal therapy with any hormonal agents such as ralozifene, Tamoxifen or other selective estrogen receptor modulators (SERMs), either for osteoporosis or prevention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada